CLINICAL TRIAL: NCT05405270
Title: Predicting Response In Cervical Intraepithelial Neoplasia to Topical Imiquimod Treatment
Acronym: PRedICT-TOPIC
Status: Recruiting | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Stichting Olijf: Dutch patient association for women with gynaecological cancer (Unknown); Leids Universitair Medisch Centrum: Department of Medical Oncology and Department of Pathology (Unknown); Maastricht Universitair Medisch Centrum: Department of Gynaecology and Department of Pathology (Unknown); Erasmus Medisch Centrum: Department of Gynaecology (Unknown); Radboud Medisch Centrum: Department of Gynaecology (Unknown)
Responsible Party: Principal Investigator, Edith van Esch, Principal Investigator, gynaecologist, Catharina Ziekenhuis Eindhoven
Other Study IDs: NL79879.100.22
Record Dates: First submitted 2022-05-19; First posted 2022-06-06 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Cervical High Grade Squamous Intraepithelial Lesion; Cervical Intraepithelial Neoplasia Grade 2/3; CIN 2/3; Cervical Intraepithelial Neoplasia
Keywords: Cervical high-grade squamous intraepithelial lesion (cHSIL); Imiquimod; Tumor immunemicroenvironment; High-risk human papilloma virus (hrHPV); Cervical intraepithelial neoplasia (CIN); Biomarker
MeSH Terms: conditions — Uterine Cervical Dysplasia | interventions — Imiquimod

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Primary cHSIL: Women with a first diagnosis of cHSIL (e.g. CIN 2 or CIN 3) who prefer treatment with imiquimod.
  Interventions: Drug: Imiquimod; Diagnostic Test: 3x vaginal swab for microbiome analysis
- Recurrent/residual cHSIL (rrcHSIL): Women who were treated for cHSIL before, but who have a residual or recurrent lesion and prefer treatment with imiquimod.
  Interventions: Drug: Imiquimod; Diagnostic Test: 3x vaginal swab for microbiome analysis
- CIN 2 observational group: Women with primary CIN 2 who prefer expectant management to await the potential of spontaneous regression.
  Interventions: Other: Expectative management; Diagnostic Test: 2x vaginal swab for microbiome analysis

INTERVENTIONS:
Drug: Imiquimod — Imiquimod 5% will be administered in the evening by either a vaginal applicator or administered on a vaginal tampon for three times a week during 16 weeks. Treatment efficacy will be evaluated after 20 weeks, by colposcopy with diagnostic biopsies, and at 6 months after completion of imiquimod therapy with cytology and if indicated histology.
  Other Names: Aldara
  Groups: Primary cHSIL; Recurrent/residual cHSIL (rrcHSIL)
Diagnostic Test: 3x vaginal swab for microbiome analysis — A vaginal swab will be taken from all patients at inclusion (before start of imiquimod), at colposcopy 20 weeks after start of imiquimod and at 6 months after completion of imiquimod treatment during follow-up appointment.
  Groups: Primary cHSIL; Recurrent/residual cHSIL (rrcHSIL)
Other: Expectative management — Expectative management of CIN 2 when preferred by the patient. Follow-up 6 months after baseline colposcopy with cytology and if indicated histology.
  Groups: CIN 2 observational group
Diagnostic Test: 2x vaginal swab for microbiome analysis — A vaginal swab will be taken from all patients at inclusion and at 6 months after inclusion during follow-up appointment.
  Groups: CIN 2 observational group

SUMMARY:
Imiquimod is a good non-invasive treatment option for women with cervical high-grade squamous intraepithelial neoplasia (cHSIL), especially those with a possible (future) pregnancy wish. Complete response to imiquimod occurs in 55-73% of patients, however side-effects of imiquimod are common and can be extensive. Therefore, biomarkers which can predict response to imiquimod therapy are warranted, to increase therapy efficacy and to avoid side effects in patients who will not respond.

This prospective, multi-center cohort study aims to validate the potential of immune related biomarkers to predict the clinical response of patients with primary cHSIL to imiquimod, aims to explore the value of these immune biomarkers in recurrent/residual cHSIL to predict treatment responses for imiquimod and aims to explore their potential in spontaneous regression of cHSIL (CIN2).

DETAILED DESCRIPTION:
RATIONALE: A persistent high risk Human Papilloma Virus (hrHPV) infection can cause (pre)malignant anogenital lesions of the cervix, vulva or vagina. Cervical high grade squamous intraepithelial lesions (cHSIL) have a malignant potential and require adequate therapy. The natural history of cHSIL is unpredictable: ~25% of cHSIL will regress, while 18% will progress to invasive cervical cancer. The standard treatment of histologically confirmed cHSIL is surgical excision by large loop excision of the transformation zone (LLETZ), with potential complications, such as hemorrhage, infection and an increased risk of preterm birth in subsequent pregnancies. Imiquimod cream has been studied as a non-invasive treatment alternative and the recent TOPIC-3 trial for cHSIL a complete response rate of 55% upon imiquimod therapy was reported. Imiquimod is now considered as a standard non-surgical therapy for patients with cHSIL in the Netherlands, especially in those patients with a future pregnancy wish. Side-effects of imiquimod therapy however are common and can be extensive, consisting mostly of local inflammation and burning, but also systemic adverse events such as headache and flu-like symptoms. Therapy adherence is challenging with up to 20% discontinuation of treatment due to the side effects and the 16 week treatment duration. As such, biomarkers which can predict response to imiquimod therapy are warranted, to increase therapy efficacy and to avoid side effects in patients who will not respond. Our previous work shows that clinical response to imiquimod in cHSIL is associated with a coordinated pre-existing type 1 T cell- and inflammatory myeloid cell infiltration and provided the first set of parameters that potentially can function together as a predictive biomarker CIBI (CHSIL Immune Biomarker for Imiquimod).

OBJECTIVE: This study aims to validate the potential of immune related biomarkers to predict the clinical response of patients with primary cHSIL to imiquimod and aims to explore the value of these immune biomarkers in recurrent/residual cHSIL to predict treatment responses for imiquimod and aims to explore their potential in spontaneous regression of cHSIL (CIN2).

STUDY DESIGN: Multicenter, real-life prospective cohort validation study.

STUDY POPULATION: We aim to include 316 women with a primary histological diagnosis of cHSIL, 50 patients with residual/recurrent histological diagnosis of cHSIL treated with imiquimod and 50 patients with cHSIL (e.g. CIN 2) not treated to await potential spontaneous regression according to the real life setting.

INTERVENTION: Patients are included in the study if they prefer imiquimod treatment, as standard care, for their cHSIL lesion or choose for expectative management of cHSIL (e.g. CIN2), according to the real-life clinical setting in the Netherlands. Patients are treated by a 16-week regime of imiquimod 5% cream, applied three times a week. Treatment efficacy will be evaluated after 20 weeks, by colposcopy with diagnostic biopsies, and at 6 months after completion of imiquimod therapy with cytology or if indicated histology. At inclusion, at 20 weeks and after 6 months a vaginal swab will be taken to evaluate the vaginal microbiome. Therapy adherence and side effects will be registered.

PRIMARY STUDY OBJECTIVES:

* Confirm the relationship between a complete clinical response to imiquimod and the increased epithelial and stromal infiltration of CD4+ T cells, CD11c+ cells and/or M1-like macrophages as well as the decreased infiltration with FoxP3+ Tregs in primary cHSIL.
* Validate the association of CIBI to a complete response to imiquimod treatment in primary cHSIL.
* Determine the sensitivity and specificity of CIBI in patients with primary cHSIL lesions to estimate the predictive value for therapy efficacy upon imiquimod treatment.

SECONDARY STUDY OBJECTIVES:

* Explore the CIBI as a predictive biomarker for therapy efficacy to imiquimod treatment in patients with residual/recurrent cHSIL (rrcHSIL).
* Explore the CIBI as a predictive biomarker for spontaneous regression of cHSIL (e.g. CIN2).
* Determine the vaginal microbiome in cHSIL patients treated with imiquimod or not treated to explore the potential interaction of the vaginal microbiome and composition of immune infiltrates in relation to imiquimod treatment and the relation to spontaneous regression.

NATURE AND EXTENT OF THE BURDEN AND RISKS ASSOCIATED WITH PARTICIPATION, BENEFIT AND GROUP RELATEDNESS: The burden associated with participation to this study is minimal since patients are included in accordance to real-life selection. If patients prefer imiquimod treatment for the therapy for their cHSIL lesion after consultation with the gynecologist they will be treated following a standard protocol, following the national guideline for cHSIL (CIN, AIS en VAIN.pdf). The burden for patients to participate in the study lies in an extra biopsy taken at colposcopy at 20 weeks and taking vaginal cultures for microbiome analysis. The benefit for the patients lies in extra support via telephonic consultation and close monitoring. For the patients in the observational arm with no treatment, no extra examinations will be performed according to the national guideline for cHSIL, only data and tissue will be used and two vaginal swabs taken. For the study cohort the benefit is limited but if we are able to identify a clinical predictive biomarker for spontaneous regression or imiquimod in cHSIL, this may increase therapy efficacy for future cHSIL patients by patient selection preventing unnecessary imiquimod therapy.

ELIGIBILITY:
Inclusion Criteria:

* Primary cHSIL lesions (e.g. CIN3 or CIN 2), histologically confirmed by diagnostic biopsy Nota bene: In case of CIN 2, expectative management must be discussed according to the Dutch national guideline with the patient, if the patient prefers imiquimod therapy the patient can be treated with imiquimod and enrolled in the study, if the patient prefers expectative management they can be enrolled in the observational CIN 2 group.
* Recurrent or residual cHSIL lesions after initial LLETZ treatment (e.g. CIN2 or CIN3), histologically confirmed by diagnostic biopsy
* Age of 18 years or older

Exclusion Criteria:

* Concomitant diagnoses of VAIN (vaginal intraepithelial neoplasia e.g. vaginal HSIL)
* PAP (Papanicolaou) 4 cytology as indication for the baseline colposcopy at study entrance
* Adenocarcinoma in situ (AIS) diagnosis
* Previous imiquimod therapy for cHSIL
* Previous cervical malignancy
* Current malignant disease
* Immunodeficiency (including HIV/AIDS and immunosuppressive medication)
* Pregnancy
* Legal incapability
* Insufficient knowledge of the Dutch language

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only patients who have a cervix uteri are eligible.
Study Population: Patients will be included in real-life outpatient clinic setting and treated according to standard Dutch therapy guidelines.
  We aim to enroll 310 patients with primary cHSIL and 50 patients with rrcHSIL treated with imiquimod and 50 cHSIL (CIN 2) patients not treated in the observational arm.
Sampling Method: Probability Sample
Enrollment: 410 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Confirm association of 'hot signature' immune infiltrates in cHSIL with complete clinical responses to imiquimod | Up to 3 years
  Confirm the relationship between a complete clinical response to imiquimod and the increased epithelial and stromal infiltration of CD4+ T cells, CD11c+ cells and/or M1-like macrophages as well as the decreased infiltration with FoxP3+ Tregs in primary cHSIL.
Validate immune biomarker CIBI for imiquimod for predicting complete response in cHSIL | Up to 3 years
  Defined as the sum of the numbers of either epithelial or stromal CD4+/CD11c+/M1+ cells per square millimeter minus the number of FoxP3+ cells per square millimeter, with a complete response to imiquimod treatment in primary cHSIL.
Determine the sensitivity and specificity of the CIBI in cHSIL | Up to 3 years
  Determine the sensitivity and specificity of the CIBI in patients with primary cHSIL lesions to estimate the predictive value for therapy efficacy upon imiquimod treatment.

SECONDARY OUTCOMES:
Explore the role of CIBI in therapy responses to imiquimod in rrcHSIL | Up to 3 years
  Explore the CIBI as a predictive biomarker for therapy efficacy to imiquimod treatment in patients with residual/recurrent cHSIL (rrcHSIL).
Explore the role of CIBI in prediction of spontaneous regression of CIN 2 | Up to 3 years
  Explore the CIBI as a predictive biomarker for spontaneous regression of cHSIL (e.g. CIN2).
Determine treatment efficacy upon imiquimod therapy. | During imiquimod treatment, 20 weeks after start of imiquimod and 6 months after completion of imiquimod treatment
  Treatment efficacy will be evaluated by determination of clinical responses at 20 weeks and at 6 months by either complete responder (CR), partial responder (PR), non-responder (NR) or progressive disease (PD) assessed by histology from biopsy and/or cytology from papsmear.
Determine therapy adherence upon imiquimod therapy. | During imiquimod treatment (16 weeks)
  Therapy adherence will be evaluated by patient reported use on the calendar by registrating the amount of imiquimod applications per week.
Determine reported side effects upon imiquimod therapy. | During imiquimod treatment (16 weeks)
  Reported side effects will be evaluated by documentation of side effects on the calendar.
Determine treatment HPV clearance upon imiquimod treatment. | Before start of imiquimod treatment, 20 weeks after start imiquimod treatment, 6 months after completion of imiquimod treatment.
  HPV clearance will be tested according to the absence or presence of hrHPV infection according to the local pathology sites via standard operating procedures.
Evaluate maintenance of lesion regression after imiquimod treatment | 24 months and 5 year follow-up with cytology and histology if necessary
  Determination of recurrent cHSIL or progression to cervical cancer.
Evaluate time to recurrence or progression of cHSIL. | 24 months and 5 year follow-up with cytology and histology if necessary
  Determination of time to recurrence or progression of cHSIL.
Explore and evaluate other potential more specific predictive (immune) biomarkers in cHSIL | Up to 3 years
  For example dedicated gene expression profiles by Nanostring and gene methylation assays.
Develop a simplified pathological scoring system | Up to 3 years
  Explorative development of a simplified dual immunohistochemistry protocol to identify the hot signature and exploration of the predictive value of this 'immunoscore' in cHSIL.
Validate the CIBI via single immunohistochemistry | Up to 3 years
  Defined as epithelial or stromal cluster of differentiation (CD) 4+/CD11c+/CD68+ cells per square millimeter with a complete response to imiquimod treatment in primary cHSIL.
Determine the vaginal microbiome in cHSIL patients | Baseline, 20 weeks after start of imiquimod and 6 months after completion of imiquimod treatment
  To explore the potential interaction of the vaginal microbiome and composition of immune infiltrates in relation to imiquimod treatment and the relation to spontaneous regression.

CONTACTS AND LOCATIONS:
Overall Officials: Edith Van Esch, MD, PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (15):
- Netherlands (15):
  - Amphia, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Tergooi MC, Hilversum
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Leiden Universitair Medisch Centrum, Leiden
  - Maastricht Universitair Medisch Centrum, Maastricht
  - Radboudumc, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
  - Franciscus Gasthuis & Vlietland, Rotterdam
  - HagaZiekenhuis, The Hague
  - Diakonessenhuis, Utrecht
  - Máxima MC, Veldhoven
  - VieCuri Medisch Centrum, Venlo
  - Isala, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] de Witte CJ, van de Sande AJ, van Beekhuizen HJ, Koeneman MM, Kruse AJ, Gerestein CG. Imiquimod in cervical, vaginal and vulvar intraepithelial neoplasia: a review. Gynecol Oncol. 2015 Nov;139(2):377-84. doi: 10.1016/j.ygyno.2015.08.018. Epub 2015 Aug 31. PMID 26335596
- [Background] Loopik DL, van Drongelen J, Bekkers RLM, Voorham QJM, Melchers WJG, Massuger LFAG, van Kemenade FJ, Siebers AG. Cervical intraepithelial neoplasia and the risk of spontaneous preterm birth: A Dutch population-based cohort study with 45,259 pregnancy outcomes. PLoS Med. 2021 Jun 4;18(6):e1003665. doi: 10.1371/journal.pmed.1003665. eCollection 2021 Jun. PMID 34086680
- [Background] Hendriks N, Koeneman MM, van de Sande AJM, Penders CGJ, Piek JMJ, Kooreman LFS, van Kuijk SMJ, Hoosemans L, Sep SJS, de Vos Van Steenwijk PJ, van Beekhuizen HJ, Slangen BFM, Nijman HW, Kruitwagen RFPM, Kruse AJ. Topical Imiquimod Treatment of High-grade Cervical Intraepithelial Neoplasia (TOPIC-3): A Nonrandomized Multicenter Study. J Immunother. 2022 Apr 1;45(3):180-186. doi: 10.1097/CJI.0000000000000414. PMID 35180719
- [Background] Abdulrahman Z, de Miranda N, van Esch EMG, de Vos van Steenwijk PJ, Nijman HW, J P Welters M, van Poelgeest MIE, van der Burg SH. Pre-existing inflammatory immune microenvironment predicts the clinical response of vulvar high-grade squamous intraepithelial lesions to therapeutic HPV16 vaccination. J Immunother Cancer. 2020 Mar;8(1):e000563. doi: 10.1136/jitc-2020-000563. PMID 32169871
- [Background] Abdulrahman Z, de Miranda NFCC, Hellebrekers BWJ, de Vos van Steenwijk PJ, van Esch EMG, van der Burg SH, van Poelgeest MIE. A pre-existing coordinated inflammatory microenvironment is associated with complete response of vulvar high-grade squamous intraepithelial lesions to different forms of immunotherapy. Int J Cancer. 2020 Nov 15;147(10):2914-2923. doi: 10.1002/ijc.33168. Epub 2020 Jul 3. PMID 32574376
- [Background] Galon J, Bruni D. Approaches to treat immune hot, altered and cold tumours with combination immunotherapies. Nat Rev Drug Discov. 2019 Mar;18(3):197-218. doi: 10.1038/s41573-018-0007-y. PMID 30610226
- [Background] Muntinga CLP, de Vos van Steenwijk PJ, Bekkers RLM, van Esch EMG. Importance of the Immune Microenvironment in the Spontaneous Regression of Cervical Squamous Intraepithelial Lesions (cSIL) and Implications for Immunotherapy. J Clin Med. 2022 Mar 5;11(5):1432. doi: 10.3390/jcm11051432. PMID 35268523
- [Background] Mitra A, MacIntyre DA, Lee YS, Smith A, Marchesi JR, Lehne B, Bhatia R, Lyons D, Paraskevaidis E, Li JV, Holmes E, Nicholson JK, Bennett PR, Kyrgiou M. Cervical intraepithelial neoplasia disease progression is associated with increased vaginal microbiome diversity. Sci Rep. 2015 Nov 17;5:16865. doi: 10.1038/srep16865. PMID 26574055
- [Background] Ovestad IT, Gudlaugsson E, Skaland I, Malpica A, Kruse AJ, Janssen EA, Baak JP. Local immune response in the microenvironment of CIN2-3 with and without spontaneous regression. Mod Pathol. 2010 Sep;23(9):1231-40. doi: 10.1038/modpathol.2010.109. Epub 2010 May 28. PMID 20512116
- [Background] Loopik DL, Bentley HA, Eijgenraam MN, IntHout J, Bekkers RLM, Bentley JR. The Natural History of Cervical Intraepithelial Neoplasia Grades 1, 2, and 3: A Systematic Review and Meta-analysis. J Low Genit Tract Dis. 2021 Jul 1;25(3):221-231. doi: 10.1097/LGT.0000000000000604. PMID 34176914